CLINICAL TRIAL: NCT01794988
Title: Can Therapy Alter CNS Processing of Chronic Pain: A Longitudinal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Magdalena Naylor, MD, PhD, Magdalena R. Naylor, MD, PhD, University of Vermont
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR059674-03 (NIH); R01AR059674-03 (NIH)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pain
Keywords: Acute Pain; Low Back Pain; Back Pain; Functional Magnetic Resonance Imaging (fMRI); Cognitive Behavioral Therapy; Pain Education
MeSH Terms: conditions — Chronic Pain; Acute Pain; Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group Cognitive Behavioral Therapy (Experimental): Participants will undergo 11 weeks of group cognitive behavioral therapy (CBT) and a pre- and post-intervention MRI brain scan.
  Interventions: Behavioral: Group Cognitive Behavioral Therapy
- Pain Education (Active Comparator): Participants will receive 11 weeks of pain education and a pre- and post-intervention MRI brain scan.
  Interventions: Behavioral: Pain Education
- Therapeutic Interactive Voice Response (Experimental): Four months of therapeutic interactive voice response (TIVR).
  Interventions: Behavioral: Therapeutic Interactive Voice Response
- No TIVR (Active Comparator): Control - no intervention
  Interventions: Behavioral: NO TIVR

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — Each CBT session will last 90 minutes and will teach participants specific skills to better cope with chronic pain. These skills will include breathing exercises, distraction, and relaxation techniques.
  Arms: Group Cognitive Behavioral Therapy
Behavioral: Pain Education — Subjects will receive mailed educational materials to their homes on a weekly basis. Weekly materials will contain information about the nature of chronic back pain, treatment options, exercises and stretching techniques for maintaining strength and flexibility, and proper protection for a healthy back. Pain education is the standard of care for most outpatient clinics.
  Arms: Pain Education
Behavioral: Therapeutic Interactive Voice Response — Therapeutic Interactive Voice Response as a daily self monitoring and relapse prevention tool with didactic reviews and practices of recorded skills and monthly feedback based on daily calls.
  Arms: Therapeutic Interactive Voice Response
Behavioral: NO TIVR — Control - no intervention
  Arms: No TIVR

SUMMARY:
The purpose of this study is to investigate whether a psycho-therapeutic approach, group Cognitive Behavioral Therapy (CBT) plus a relapse prevention program, Therapeutic Interactive Voice Response (TIVR), modifies the dysfunctional sensory, emotional, and cognitive neural circuitry associated with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months of muscular-skeletal, non-neuropathic pain

Exclusion Criteria:

* Malignancy causing or influencing chronic pain
* Radiation or chemotherapy, or metastatic cancer of any type
* Reflex Sympathetic Dystrophy (RSD) and/or neuropathic pain
* Neurological disorders such as epilepsy or stroke, or other medical conditions
* Psychiatric disorders
* Opioid medication use for pain management
* Past year history of illicit drug use that can result in altered cognition
* Pregnancy
* Exceeding weight limit of the MRI scanner
* Incompatible implants due to MRI safety
* Awaiting pain related surgical procedure
* Involved in pain-related litigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Pain | Seven Months

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Naylor, MD, PhD, Principal Investigator — Faculty, University of Vermont College of Medicine
Locations (1):
- University of Vermont College of Medicine, MindBody Medicine Clinic, Burlington, Vermont, United States

REFERENCES:
- See also: MindBody Medicine Clinic Chronic Pain Research — http://www.uvm.edu/~mbmc/?Page=research/chronicPain.html&SM=researchSM.html